CLINICAL TRIAL: NCT01262508
Title: Development of Algorithms to Detect and Predict Hemodynamic Instability in Patients at Risk
Brief Title: Development of Algorithms to Predict Hemodynamic Instability
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie Christian Meyer, MD, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: Autonomics - Prediction
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Sudden Cardiac Death
Keywords: autonomic nervous system
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Risk Population: Patients being suspected to be at risk of hemodynamic instability due to medical history

SUMMARY:
Hemodynamic monitoring in hospitalized patients is crucial since in clinical practice unexpected deterioration of cardiovascular function remains a serious problem and an important cause of death. Novel perspectives in reflex testing of the autonomic nervous system might be useful to protect some patients from cardiovascular events by detecting cardiovascular deteriorations. In addition, standard pulse oximetry in low acuity settings is nowadays predominately used to monitor peripheral oxygen saturation. Of note, there is evidence that additional analyses of pulse wave characteristics might be a valuable source of information to generate additional insights into the cardiorespiratory status of the patient. Herein, we aim to develop novel algorithms in order to protect in-hospital patients from cardiovascular events in consequence of hemodynamic instability in the future.

DETAILED DESCRIPTION:
70 datasets from hospitalized patients will be acquired in order to characterize the functional status of the autonomic nervous system as well as hemodynamics during baseline and during standard procedures including physical exercise testing and head-up tilt table testing.

Autonomic reflex testing:

* Heart Rate Characteristics
* Heart Rate Variability
* Heart Rate Turbulence
* Blood Pressure Variability
* Baroreflex Sensitivity
* Hyperoxic Chemoreflex Sensitivity

Hemodynamic Monitoring:

* Heart Rate Trends
* Blood Pressure Trends
* Pulse Wave Characteristics
* Cardiac Output
* Peripheral Vascular Resistance
* Context information

ELIGIBILITY:
Inclusion Criteria:

* hospitalization
* Age > 17 years

Exclusion Criteria:

* documented diseases of the central nervous system
* impairment of mental health
* age > 85 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients being at risk of sudden cardiac death
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Autonomic Dysfunction | 24 hours
  Dysfunction of the autonomic nervous system as assessed by autonomic reflex testing

SECONDARY OUTCOMES:
Hemodynamic Deterioration | 24 hours
  Acute hemodynamic changes (Blood pressure changes > 10 mm Hg, heart rate changes > 5 bpm both within 30 seconds) of a patient as assessed by hemodynamic monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, Study Chair — University of Duesseldorf; Malte Kelm, MD, PhD, Study Director — University of Duesseldorf
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Jungen C, Zeus T, Balzer J, Eickholt C, Petersen M, Kehmeier E, Veulemans V, Kelm M, Willems S, Meyer C. Left Atrial Appendage Closure Guided by Integrated Echocardiography and Fluoroscopy Imaging Reduces Radiation Exposure. PLoS One. 2015 Oct 14;10(10):e0140386. doi: 10.1371/journal.pone.0140386. eCollection 2015. PMID 26465747
- [Derived] Drexel T, Eickholt C, Muhlsteff J, Ritz A, Siekiera M, Kirmanoglou K, Schulze V, Shin DI, Balzer J, Rassaf T, Kelm M, Meyer C. Vagal heart rate control in patients with atrial fibrillation: impact of tonic activation of peripheral chemosensory function in heart failure. Adv Exp Med Biol. 2013;755:287-97. doi: 10.1007/978-94-007-4546-9_37. PMID 22826079
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie